CLINICAL TRIAL: NCT02777983
Title: Brief Mobile Education at the Point of Care to Influence Healthcare Decisions Related Low Back Pain Management in Primary Care
Brief Title: MOBile Instruction for Low Back Pain (MOBIL)
Acronym: MOBIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Rhon, Director of Physical Therapy, Center for the Intrepid, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2015.029
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Low Back Pain
Keywords: patient education; low back pain; technology
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education Group (Experimental): This will consist of a 6-minute educational video app created and delivered within an application (mobile app) that will be interactive in nature, asking multiple-choice questions at the end to help reinforce key points of the video message. It will include self-management guidance based on evidence related to activity, exercise, and other behavioral components known to influence the prognosis of low back pain. Subjects will also receive the 1-page general conditioning handout that the usual care group will receive.
  Interventions: Behavioral: Educational Video App
- Usual Care Group (No Intervention): Subjects randomized to usual care will receive a 1-page generic informational handout on general conditioning recommended for low back pain, in addition to whatever education the subject's PCP decides to provide.

INTERVENTIONS:
Behavioral: Educational Video App — The content of the app will be grounded in a biopsychosocial model and modeled on the Back Book, a booklet developed to help modify beliefs and behavior of patients with LBP. Essentially this will take the primary concepts and ideas often given in print or verbal form, and present it in a more engaging and dynamic fashion.
  Other Names: Mobile Technology Education
  Arms: Education Group

SUMMARY:
The purpose of this project is to measure the impact of a short educational session on outcomes for patients consulting in primary care for low back pain. Subjects will be patients consulting to their primary care provider for a primary complaint and new episode of low back pain. Subjects will be randomized to receiving the educational tool versus usual care (information only without an educational component) in the clinic immediately prior to seeing their PCP. Patients will be followed for a 6-month period, and outcome measures will be collected and compared across both groups.

DETAILED DESCRIPTION:
Patients that arrive for an initial evaluation for low back pain will be randomized to either receive the video education via an application (app) on a tablet computer, or usual care (which consists of information in the form of a handout but no further education prior to seeing the Primary Care Provider - PCP). To control for exposure to the tablet computer, subjects in both groups will use the tablet computer to fill out the self-reported outcome measures.

This will all take place while the patient is waiting to see their PCP, who will be blinded to the educational intervention that the patient received. After enrollment and completion of baseline outcome measures and surveys, the subject will be randomized to one of the 2 arms, receive the intervention, and then proceed to have their appointment with their PCP. The appointment with the PCP will proceed per usual care standards, with no additional research interventions. The subjects will be contacted for a follow-up at 1 and 6 months for assessment of self-reported outcomes measuring pain, function, and disability. The investigators will also abstract healthcare utilization from claims data and compare variables of healthcare use between both groups over the 6-month period following enrollment (radiographs, MRIs, prescription opioids, and specialty referrals).

ELIGIBILITY:
Inclusion Criteria:

1. A Tricare beneficiary with a primary complaint of low back pain consulting in a primary care clinic
2. Between the age of 18 - 50 years
3. Read and speak English well enough to interact with the mobile education technology, provide informed consent and follow study instructions

Exclusion Criteria:

1. History of prior surgery to the lumbosacral spine
2. Medical "red flags" of a potentially serious condition including cauda equina syndrome, major or rapidly progressing neurological deficit, fracture, cancer, infection, or systemic disease
3. Known current pregnancy or history of pregnancy in the last 6 months
4. Already seen in primary care for an episode of low back pain within the last 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Healthcare Utilization | 6 months
  This will include an a frequency count of diagnostic imaging orders and types, specialty referrals, and medication use (primarily prescription opiates).

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System 29 Item Subscale (PROMIS-29) | 0, 1, 6 months
  The PROMIS 29-item short form efficiently assesses several outcomes important to patients with a neuromusculoskeletal injury, including pain intensity and interference, sleep disturbance, anxiety, depression, fatigue, and social role participation using items developed with rigorous methodology and patient input. The PROMIS-29 scores have been found valid for patients with orthopedic injuries with minimal clinically important change thresholds of 2-4 points for most scales. It has also been used to successfully measure psychosocial resiliency in patients with disability.
Keele STarT Back Screening Tool (SBST) | 0, 1, 6 months
  The Keele STarT Back Screening Tool classifies patients into one of three risk categories (low, medium, and high) for targeted treatment, based on the presence of potentially modifiable physical and psychological prognostic indicators for persistent, disabling symptoms, identified through 9 questions. Patients are classified as "low risk" of future disabling LBP if they score positively on fewer than 4 questions. The remainder are then subdivided into "medium risk" (physical and psychosocial indicators for poor outcome, but without high levels of psychological indicators) and "high risk" (high levels of psychological prognostic indicators with or without physical indicators).
Optimal Screening for Prediction of Referral and Outcome Yellow Flags assessment tool (OSPRO-YF) | 0, 1, 6 months
  Measures of psychosocial risk factors taken early after injury and sequentially over time represent an important and relevant clinical necessity, as psychosocial risk factors can vary over time. Some preliminary work on how sequential assessment may improve predictive capabilities has been performed. In previous studies of the SBST, baseline risk status was compared to prediction from 4-week risk status, and 4-week change in risk status for prediction of 6 month pain and disability outcomes following low back pain. The results indicated that prediction improved when 4-week risk status or 4-week change in risk status was incorporated into predictive models. In particular, those with worsened 4 week change in psychosocial risk status (i.e. increasing pain associated distress) had notably worse 6 month outcomes. This provides promising preliminary data for investigating how these change patterns influence patient outcomes in patients with low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rhon, DPT, DSc, Principal Investigator — Brooke Army Medical Center; Baylor University
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for data must go through a Data Sharing Agreement Application submitted and approved through the Defense Health Agency
Time Frame: DHA usually approves Data Sharing Agreements for up to 1 year at a time
Access Criteria: Requires a Data Sharing Agreement Application to be submitted through the US Defense Health Agency
URL: https://www.health.mil/Military-Health-Topics/Privacy-and-Civil-Liberties/Submit-a-Data-Sharing-Application

REFERENCES:
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] George SZ, Childs JD, Teyhen DS, Wu SS, Wright AC, Dugan JL, Robinson ME. Brief psychosocial education, not core stabilization, reduced incidence of low back pain: results from the Prevention of Low Back Pain in the Military (POLM) cluster randomized trial. BMC Med. 2011 Nov 29;9:128. doi: 10.1186/1741-7015-9-128. PMID 22126534
- [Background] Darlow B, Fullen BM, Dean S, Hurley DA, Baxter GD, Dowell A. The association between health care professional attitudes and beliefs and the attitudes and beliefs, clinical management, and outcomes of patients with low back pain: a systematic review. Eur J Pain. 2012 Jan;16(1):3-17. doi: 10.1016/j.ejpain.2011.06.006. PMID 21719329
- [Background] Foster NE, Delitto A. Embedding psychosocial perspectives within clinical management of low back pain: integration of psychosocially informed management principles into physical therapist practice--challenges and opportunities. Phys Ther. 2011 May;91(5):790-803. doi: 10.2522/ptj.20100326. Epub 2011 Mar 30. PMID 21451095
- [Background] Godges JJ, Anger MA, Zimmerman G, Delitto A. Effects of education on return-to-work status for people with fear-avoidance beliefs and acute low back pain. Phys Ther. 2008 Feb;88(2):231-9. doi: 10.2522/ptj.20050121. Epub 2007 Dec 4. PMID 18056753
- [Background] Burton AK, Waddell G, Tillotson KM, Summerton N. Information and advice to patients with back pain can have a positive effect. A randomized controlled trial of a novel educational booklet in primary care. Spine (Phila Pa 1976). 1999 Dec 1;24(23):2484-91. doi: 10.1097/00007632-199912010-00010. PMID 10626311
- [Background] Cherkin D, Deyo RA, Berg AO. Evaluation of a physician education intervention to improve primary care for low-back pain. II. Impact on patients. Spine (Phila Pa 1976). 1991 Oct;16(10):1173-8. doi: 10.1097/00007632-199110000-00008. PMID 1836677
- [Background] Moore JE, Von Korff M, Cherkin D, Saunders K, Lorig K. A randomized trial of a cognitive-behavioral program for enhancing back pain self care in a primary care setting. Pain. 2000 Nov;88(2):145-153. doi: 10.1016/S0304-3959(00)00314-6. PMID 11050369
- [Derived] Rhon DI, Mayhew RJ, Greenlee TA, Fritz JM. The influence of a MOBile-based video Instruction for Low back pain (MOBIL) on initial care decisions made by primary care providers: a randomized controlled trial. BMC Fam Pract. 2021 Oct 9;22(1):200. doi: 10.1186/s12875-021-01549-y. PMID 34627152